CLINICAL TRIAL: NCT04399720
Title: Root Canal Treatment of Compromised Teeth as Alternative Treatment in Patients Under Bisphosphonate Therapy: 60-month Results of a Prospective Clinical Study
Brief Title: Root Canal Treatment Outcome in Patients Under Bisphosphonate Therapy
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Fausto Zamparini, DDS,MS,PhD, University of Bologna
Other Study IDs: bifosfonendo
Record Dates: First submitted 2020-05-20; First posted 2020-05-22 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Root Canal Infection; Bisphosphonate-Associated Osteonecrosis; Periapical Abscess; Endodontically Treated Teeth
Keywords: success rate; survival rate; endodontic treatment
MeSH Terms: conditions — Bisphosphonate-Associated Osteonecrosis of the Jaw; Periapical Abscess; Tooth, Nonvital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BPS group: patients under Bisphosphonate therapy for at least 24 months
  Interventions: Procedure: Root canal treatment
- healthy patients: healthy patients not assuming with no previous Bisphosphonate assumption
  Interventions: Procedure: Root canal treatment

INTERVENTIONS:
Procedure: Root canal treatment — Root canal treatment using a standard manual k file instrumentation and carrier-based root canal filling technique

SUMMARY:
The aim of this study was to evaluate the survival rate and healing time of compromised teeth and seriously compromised teeth that were endodontically treated in patients which received bisphosphonate therapy . Clinical complications, success and survival rate was reported. Mean clinical parameters, clinical symptoms and presence of periapical radilucency were recorded.

DETAILED DESCRIPTION:
The study was conducted in one University Endodontic Clinical Department - Dental School between January 2009 and December 2017.

Root canal treatment was performed according previously reported operative protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by endodontic disease and able to attend a hygiene recall program

Exclusion Criteria:

* inability to attend a recall hygien program

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Similar geographic provenience
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2009-01-07 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
health patients | 5 years
  assessment of periapical index (PAI)

SECONDARY OUTCOMES:
Complications | 5 years
  extraction periapical re exacerbation during before the endline ( 5 years)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pirani C, Chersoni S, Montebugnoli L, Prati C. Long-term outcome of non-surgical root canal treatment: a retrospective analysis. Odontology. 2015 May;103(2):185-93. doi: 10.1007/s10266-014-0159-0. Epub 2014 Jun 8. PMID 24908421
- [Result] Prati C, Pirani C, Zamparini F, Gatto MR, Gandolfi MG. A 20-year historical prospective cohort study of root canal treatments. A Multilevel analysis. Int Endod J. 2018 Sep;51(9):955-968. doi: 10.1111/iej.12908. Epub 2018 Mar 7. PMID 29432651